CLINICAL TRIAL: NCT05745350
Title: An Open-Label, Single-Arm, Phase II Study of Pembrolizumab, Plinabulin Plus Etoposide and Platinum as First-Line Therapy for Extensive-Stage Small-Cell Lung Cancer
Brief Title: First Line Pembrolizumab, Plinabulin Plus Etoposide and Platinum (EP) for ES-SCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xiaorong Dong (Other)
Responsible Party: Sponsor-Investigator, Xiaorong Dong, Principal Investigator, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Organization: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KeyPemls-005
Record Dates: First submitted 2023-02-05; First posted 2023-02-27 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Small Cell Lung Cancer Extensive Stage
MeSH Terms: interventions — pembrolizumab; NPI 2358; Etoposide; Platinum

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: Pembrolizumab, Plinabulin plus Etoposide and Platinum

INTERVENTIONS:
Drug: Pembrolizumab, Plinabulin plus Etoposide and Platinum — Pembrolizumab 200 mg IV every 3 weeks (Q3W) on Day 1; Etoposide 100 mg/m2 IV Q3W on Days 1, 2, and 3; Carboplatin AUC 5 IV Q3W on Day 1 or Cisplatin 75 mg/m2 IV Q3W on Day 1; Plinabulin 30mg/m2 IV Q3W on Day 1.

SUMMARY:
Monoclonal antibodies against programmed death 1 (PD-1) and its ligand PD-L1 have shown efficacy in patients with ES-SCLC in the monotherapy and combination therapy settings. Up to now, Atezolizumab and Durvalumab has been approved for first line treatment for ES-SCLC in China combined with EP or EC. Besides, KEYNOTE-604 study revealed that adding pembrolizumab to standard first-line EP significantly improves PFS in patients with ES-SCLC and is associated with durable responses in a subset of patients. 12-m PFS rate were 13.6% with pembrolizumab plus EP and 3.1% with placebo plus EP. The statistical threshold for declaring significant prolongation of OS was narrowly missed. Considering sicker pts was enrolled and the interim analysis was quite often, even though the investigators narrowly missed the OS endpoint, longer numerical OS data was observed. The latest version of NCCN SCLC guidelines still recommended pembrolizumab as an option for ES-SCLC patients.

Plinabulin received breakthrough designation from both US and China FDA for CIN (Chemotherapy Induced Neutropenia) prevention indication. As a "pipeline in a drug," plinabulin is being broadly studied in combination with various immuno-oncology agents that could boost the effects of the PD-1/PD-L1 antibodies and re-sensitize PD-1/PD-L1 antibody resistant patients. In a poster released at 2021 ASCO conference, a phase I trial of Plinabulin in combination with nivolumab and ipilimumab in patients with relapsed small cell lung cancer: Big Ten Center Research Consortium (BTCRC-LUN17-127) study. Plinabulin in combination with nivolumab and ipilimumab was safe and well tolerated with promising efficacy signal of 46% ORR.

From above, Pembrolizumab, Plinabulin plus Etoposide and Platinum as First-Line Therapy for ES-SCLC should be a promising combination therapy, as the investigators expect increased efficacy and reduced toxicity with the addition of Plinabulin. In this proof of concept phase II study, the investigators will investigate that the efficacy and safety of Pembrolizumab, Plinabulin plus Etoposide and Platinum as First-Line Therapy for ES-SCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Have a documented new diagnosis of SCLC by histology or cytology from brushing, washing, or needle aspiration of a defined lesion.
2. Have extensive stage disease defined as Stage IV (T any, N any, M 1a/b) by the American Joint Committee on Cancer, Eighth Edition.
3. Have at least 1 lesion that meets the criteria for being measurable, as defined by RECIST 1.1, and is appropriate for selection as a target lesion, as determined by local site investigator/radiology review.
4. Life expectancy ≥3 months.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
6. Male/female participants who are at least 18 years of age on the day of signing informed consent.
7. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
8. Have adequate organ function.
9. Criteria for known Hepatitis B and C positive subjects 9.1 Hepatitis B positive subjects

   * Participants who are HBsAg positive are eligible if they have received HBV antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to treatment.
   * Participants should remain on anti-viral therapy throughout study intervention and follow local guidelines for HBV anti-viral therapy post completion of study intervention.

   9.2 Participants with history of HCV infection are eligible if HCV viral load is undetectable at screening. Participants must have completed curative anti-viral therapy at least 4 weeks prior to the first treatment.
10. Male participants:

    A male participant must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 180 days after the last dose of study treatment and refrain from donating sperm during this period.
11. A female participant is eligible to participate if she is not pregnant, not breastfeeding.

Exclusion Criteria:

1. Has received prior systemic therapy for the treatment of SCLC.
2. Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
3. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment for another health-related problem.
4. Is expected to require any other form of antineoplastic therapy for SCLC, including radiation therapy, while on study.

   Note: Patients with PR or CR will be offered PCI therapy at the investigator's consideration at the completion of the 4 cycles of chemotherapy with pembrolizumab
5. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
6. Has had major surgery within 3 weeks prior to receiving the first dose of trial treatment or has not recovered adequately from toxicity and/or complications from an intervention prior to receiving the first dose of study treatment
7. Has active autoimmune disease that has required systemic treatment in the past 2 years (ie, with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
8. Has symptomatic ascites, pleural effusion, or pericardial effusion. A participant who is clinically stable following treatment for these conditions (including therapeutic thoraco or paracentesis) is eligible.
9. Known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ, excluding carcinoma in situ of the bladder, that have undergone potentially curative therapy are not excluded.
10. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.

    Has severe hypersensitivity (≥Grade 3) to plinabulin and/or any of its excipients.
11. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
12. Has a known history of Human Immunodeficiency Virus (HIV) infection.
13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
14. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another co-inhibitory T-cell receptor (ie, CTLA-4, OX-40, CD137) or has previously participated in a MSD pembrolizumab (MK-3475) clinical trial and Beyond Spring Plinabulin clinical trial.
15. Has had an allogenic tissue/solid organ transplant.
16. Has received a live vaccine within 30 days prior to the first dose of trial drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
17. Has a known history of active TB (Bacillus Tuberculosis).
18. Any medical conditions that in the Investigator's opinion, would impose excessive risk to the patient. Examples of such conditions include uncontrolled diabetes, infection requiring parenteral anti-infective treatment, liver failure, any altered mental status or any psychiatric condition that would interfere with the understanding of the ICF.
19. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 180 days after the last dose of trial treatment.
20. Active uncontrolled bacterial, viral, or fungal infection requiring systemic therapy.
21. Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
12-m PFS rate | From date of the first treatment to the first documented disease progression, assessed up to 24 months.
  Progression-free survival is defined as the time from the first treatment to the first documented disease progression per RECIST 1.1.

SECONDARY OUTCOMES:
ORR | up to 24 months.
  Objective response rate is defined as the proportion of subjects who have a CR or a PR.
DoR | up to 24 months.
  Time from the first assessment of CR or PR to the first assessment of PD or death.
PFS | From date of the first treatment to the first documented disease progression, assessed up to 24 months.
  Progression-free survival is defined as the time from the first treatment to the first documented disease progression.
OS | From date of the first treatment to death due to any cause, assessed up to 24 months.
  Overall survival is defined as the time from the first treatment to death due to any cause.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | up to 24 months.
  Description of characteristics and frequency of AEs.

OTHER OUTCOMES:
Exploratory Biomarker Research | up to 24 months.
  Blood and/or Tissue being collected in the study will be used to conduct a biomarker analysis study.

CONTACTS AND LOCATIONS:
Locations (1):
- Union hospital, Wuhan, Hubei, China